CLINICAL TRIAL: NCT00303745
Title: Randomized Study of Second-Line Therapy Comprising Irinotecan With or Without Capecitabine in Patients Aged At Least 75 Years With Colorectal Cancer
Brief Title: Irinotecan With or Without Capecitabine as Second-Line Therapy in Treating Older Patients With Progressive, Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453857; FFCD-0305; EU-20545; EUDRACT-2004-004742-40
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2006-12

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Irinotecan

INTERVENTIONS:
Drug: capecitabine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether irinotecan and capecitabine are more effective than irinotecan alone in treating colorectal cancer.

PURPOSE: This randomized phase II trial is studying irinotecan and capecitabine to see how well they work as second-line therapy compared to irinotecan alone in treating older patients with progressive, metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the objective response or stable disease rate in elderly patients with unresectable, progressive, metastatic colorectal cancer treated with irinotecan hydrochloride with vs without capecitabine.

Secondary

* Compare the tolerability of these regimens in these patients.
* Compare the quality of life and ability to maintain self-sufficiency of patients treated with these regimens.
* Compare the progression-free and overall survival of patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to participating center, WHO performance status (0 or 1 vs 2), number of associated comorbidities (Charlson index 0-2 vs > 2), and age (75-79 vs ≥ 80). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 2 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral capecitabine on days 1-14 and irinotecan hydrochloride IV over 90 minutes on day 1. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 12 weeks thereafter.

After completion of study therapy, patients are followed every 12 weeks.

PROJECTED ACCRUAL: A total of 78 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum

  * Unresectable disease
  * Documented progressive disease during first-line/palliative chemotherapy
* Measurable disease ≥ 1 cm that is outside prior radiation field
* No brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* No contraindication to chemotherapy
* Creatinine clearance ≥ 40 mL/min
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Alkaline phosphatase ≤ 3 times normal (5 times normal if hepatic involvement)
* Bilirubin ≤ 1.5 times normal
* Transaminases ≤ 5 times normal
* No symptomatic coronary disease or cardiac insufficiency
* No enteropathy or chronic diarrhea
* No unresolved intestinal occlusion or subocclusion
* No history of severe unexpected reaction to a fluoropyrimidine
* No other active malignancy in the past 2 years
* No hypersensitivity to irinotecan hydrochloride or its excipients
* No hypersensitivity to capecitabine or fluorouracil

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior extensive resection
* No concurrent sorivudine or similar analogs (e.g., brivudine)
* No other concurrent anticancer therapy
* Concurrent radiotherapy allowed for nontarget lesions

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
Objective response
Stable disease rate

SECONDARY OUTCOMES:
Tolerability
Quality of life
Progression-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mitry, MD, PhD — Hopital Ambroise Pare; Thomas Aparicio, Study Chair — Hopital Bichat - Claude Bernard
Locations (23):
- France (23):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Centre Hospitalier Universitaire Ambroise Pare - Boulogne, Boulogne
  - Centre Hospitalier, Chalon-sur-Saône
  - Hopital Antoine Beclere, Clamart
  - Hopital Du Bocage, Dijon
  - Clinique Pasteur, Guilherand-Granges
  - CMC Les Ormeaux, Le Havre
  - C. H. Du Mans, Le Mans
  - Hopital Robert Boulin, Libourne
  - Polyclinique des Quatre Pavillons, Lormont
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Hopital Sebastopol, C.H.U. de Reims, Reims
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - C.H. Senlis, Senlis
  - CHRU de Tours - Hopital Trousseau, Tours
  - Centre Hospitalier General - St. Nicolas, Verdun